CLINICAL TRIAL: NCT06696027
Title: Investigating the Role of Hematopoietic Mutations and Mosaic Mutation in the Y Chromosome in Autoimmune Rheumatologic Diseases
Brief Title: AYLo - AutoimmunitY and Loss of y
Acronym: AYLo
Status: Recruiting | Type: Observational
Sponsor: University of Bonn (Other)
Responsible Party: Principal Investigator, Valentin Schäfer, Principal Investigator, University Hospital, Bonn
Other Study IDs: 2024-471-BO
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Giant Cell Arteritis (GCA); Polymyalgia Rheumatica (PMR); ANCA Associated Vasculitis (AAV); Idiopathic Inflammatory Myopathies; IgG4-Related Diseases; Rheumatoid Arthritis (RA); Psoriatic Arthritis (PsA); Connective Tissue Disease; Sarcoidosis; Interstitial Lung Disease Due to Systemic Disease (Disorder); Interstitial Lung Disease (ILD); Asthma Bronchiale; COPD
Keywords: Autoimmune Diseases; Vasculitis; Large Vessel Vasculitis; Giant Cell Arteritis; Polymyalgia Rheumatica; ANCA Associated Vasculitis; Idiopathic Inflammatory Myopathies; IgG4-Related Diseases; Rheumatoid Arthritis; Psoriatic Arthritis; Connective Tissue Disease; Sarcoidosis; Interstitial Lung Disease
MeSH Terms: conditions — Giant Cell Arteritis; Polymyalgia Rheumatica; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Myositis; Immunoglobulin G4-Related Disease; Arthritis, Rheumatoid; Arthritis, Psoriatic; Connective Tissue Diseases; Sarcoidosis; Lung Diseases, Interstitial; Pulmonary Disease, Chronic Obstructive; Autoimmune Diseases; Vasculitis | interventions — Polymorphism, Single Nucleotide; Flow Cytometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood, Pax Tubes, Serum, PBMC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (13):
- Giant Cell Arteritis (GCA): Patients with GCA (cross sectional, newly diagnosed with follow-up after twelve months).
  Interventions: Diagnostic Test: Single nucleotide polymorphisms (SNP); Diagnostic Test: 3'mRNA sequencing; Diagnostic Test: Enzyme-linked immunosorbent assay (ELISA) and Legendplex Array; Diagnostic Test: Flow Cytometry; Diagnostic Test: Laboratory assessment
- Polymyalgia Rheumatica (PMR): Patients with PMR (cross sectional, newly diagnosed with follow-up after twelve months).
  Interventions: Diagnostic Test: Single nucleotide polymorphisms (SNP); Diagnostic Test: 3'mRNA sequencing; Diagnostic Test: Enzyme-linked immunosorbent assay (ELISA) and Legendplex Array; Diagnostic Test: Flow Cytometry; Diagnostic Test: Laboratory assessment
- ANCA Associated Vasculitis (AAV): Patients with AAV (cross sectional, newly diagnosed with follow-up after twelve months).
  Interventions: Diagnostic Test: Single nucleotide polymorphisms (SNP); Diagnostic Test: 3'mRNA sequencing; Diagnostic Test: Enzyme-linked immunosorbent assay (ELISA) and Legendplex Array; Diagnostic Test: Flow Cytometry; Diagnostic Test: Laboratory assessment; Diagnostic Test: Assessment of Pulmonary Involvement
- IgG4 Related Diseases: Patients with IgG4 Related Diseases (cross sectional, newly diagnosed with follow-up after twelve months).
  Interventions: Diagnostic Test: Single nucleotide polymorphisms (SNP); Diagnostic Test: 3'mRNA sequencing; Diagnostic Test: Enzyme-linked immunosorbent assay (ELISA) and Legendplex Array; Diagnostic Test: Flow Cytometry; Diagnostic Test: Laboratory assessment
- Idiopathic Inflammatory Myopathies (IIM): Patients with IIM (cross sectional, newly diagnosed with follow-up after twelve months).
  Interventions: Diagnostic Test: Single nucleotide polymorphisms (SNP); Diagnostic Test: 3'mRNA sequencing; Diagnostic Test: Enzyme-linked immunosorbent assay (ELISA) and Legendplex Array; Diagnostic Test: Flow Cytometry; Diagnostic Test: Laboratory assessment; Diagnostic Test: Assessment of Pulmonary Involvement
- Rheumatoid Arthritis (RA): Patients with RA (cross sectional, newly diagnosed with follow-up after twelve months).
  Interventions: Diagnostic Test: Single nucleotide polymorphisms (SNP); Diagnostic Test: 3'mRNA sequencing; Diagnostic Test: Enzyme-linked immunosorbent assay (ELISA) and Legendplex Array; Diagnostic Test: Flow Cytometry; Diagnostic Test: Laboratory assessment; Diagnostic Test: Assessment of Pulmonary Involvement
- Psoriatic Arthritis (PsA): Patients with PsA (cross sectional, newly diagnosed with follow-up after twelve months).
  Interventions: Diagnostic Test: Single nucleotide polymorphisms (SNP); Diagnostic Test: 3'mRNA sequencing; Diagnostic Test: Enzyme-linked immunosorbent assay (ELISA) and Legendplex Array; Diagnostic Test: Flow Cytometry; Diagnostic Test: Laboratory assessment; Diagnostic Test: Assessment of Pulmonary Involvement
- Connective Tissue Diseases (CTD): Patients with CTD (cross sectional, newly diagnosed with follow-up after twelve months).
  Interventions: Diagnostic Test: Single nucleotide polymorphisms (SNP); Diagnostic Test: 3'mRNA sequencing; Diagnostic Test: Enzyme-linked immunosorbent assay (ELISA) and Legendplex Array; Diagnostic Test: Flow Cytometry; Diagnostic Test: Laboratory assessment; Diagnostic Test: Assessment of Pulmonary Involvement
- Sarcoidosis: Patients with sarcoidosis (cross sectional, newly diagnosed with follow-up after twelve months).
  Interventions: Diagnostic Test: Single nucleotide polymorphisms (SNP); Diagnostic Test: 3'mRNA sequencing; Diagnostic Test: Enzyme-linked immunosorbent assay (ELISA) and Legendplex Array; Diagnostic Test: Flow Cytometry; Diagnostic Test: Laboratory assessment; Diagnostic Test: Assessment of Pulmonary Involvement
- Interstitial Lung Diseases (ILD): Patients with ILD (cross sectional, newly diagnosed with follow-up after twelve months).
  Interventions: Diagnostic Test: Single nucleotide polymorphisms (SNP); Diagnostic Test: 3'mRNA sequencing; Diagnostic Test: Enzyme-linked immunosorbent assay (ELISA) and Legendplex Array; Diagnostic Test: Flow Cytometry; Diagnostic Test: Laboratory assessment; Diagnostic Test: Assessment of Pulmonary Involvement
- Chronic Obstructive Pulmonary Disease (COPD): Patients with COPD (cross sectional, newly diagnosed with follow-up after twelve months).
  Interventions: Diagnostic Test: Single nucleotide polymorphisms (SNP); Diagnostic Test: 3'mRNA sequencing; Diagnostic Test: Enzyme-linked immunosorbent assay (ELISA) and Legendplex Array; Diagnostic Test: Flow Cytometry; Diagnostic Test: Laboratory assessment; Diagnostic Test: Assessment of Pulmonary Involvement
- Asthma Bronchiale: Patients with asthma bronchiale (cross sectional, newly diagnosed with follow-up after twelve months).
  Interventions: Diagnostic Test: Single nucleotide polymorphisms (SNP); Diagnostic Test: 3'mRNA sequencing; Diagnostic Test: Enzyme-linked immunosorbent assay (ELISA) and Legendplex Array; Diagnostic Test: Flow Cytometry; Diagnostic Test: Laboratory assessment; Diagnostic Test: Assessment of Pulmonary Involvement
- Healthy Control Group: Age-/ gender matched healthy controls
  Interventions: Diagnostic Test: Single nucleotide polymorphisms (SNP); Diagnostic Test: 3'mRNA sequencing; Diagnostic Test: Enzyme-linked immunosorbent assay (ELISA) and Legendplex Array; Diagnostic Test: Flow Cytometry; Diagnostic Test: Laboratory assessment; Diagnostic Test: Assessment of Pulmonary Involvement

INTERVENTIONS:
Diagnostic Test: Single nucleotide polymorphisms (SNP) — Utilizing single nucleotide polymorphisms (SNP) genotyping mosaic loss of y (mLOY) of individual patient will be assessed.
Diagnostic Test: 3'mRNA sequencing — 3'mRNA sequencing analyzes gene expression profiles related to the immune response in different study cohorts, aiding in understanding the genetic underpinnings of inflammation and its association with mLOY.
Diagnostic Test: Enzyme-linked immunosorbent assay (ELISA) and Legendplex Array — Used to measure cytokine levels in the serum of investigated patients, aiding in profiling inflammatory markers that are indicative of disease activity, response to treatment and consequence of mLOY..
Diagnostic Test: Flow Cytometry — Employed to analyze immune cell phenotypes in investigated cohorts. This test helps identify various immune cell subsets and their activation states, which are critical for understanding disease mechanisms and its association with mLOY.
Diagnostic Test: Laboratory assessment — Serum Chemistry
Diagnostic Test: Assessment of Pulmonary Involvement — Results of routine clinical assessment of pulmonary involvement (such as lung ultrasound, computed tomography, chest x-ray, whole-body plethysmography) will be compared to mLOY, ELISA/ Legendplex/ flow cytometry/ transcriptome analysis results.
  Groups: ANCA Associated Vasculitis (AAV); Asthma Bronchiale; Chronic Obstructive Pulmonary Disease (COPD); Connective Tissue Diseases (CTD); Healthy Control Group; Idiopathic Inflammatory Myopathies (IIM); Interstitial Lung Diseases (ILD); Psoriatic Arthritis (PsA); Rheumatoid Arthritis (RA); Sarcoidosis

SUMMARY:
The AYLo study (AutoimmunitY and Loss of y - Investigating the Role of Hematopoietic Mutations and Mosaic Mutation in the Y Chromosome in Autoimmune Rheumatologic Diseases) aims to systematically investigate hematopoietic mutations, such as hematopoietic (mosaic) loss of the Y chromosome (mLOY), focusing on their underlying causes, pathophysiological significance, patterns of manifestation, and impact on disease progression in autoimmune, rheumatologic disorders. This research seeks to bridge existing knowledge gaps by exploring how such mutations influence immune homeostasis, cellular function, and susceptibility to inflammation-driven pathologies.

Through the integration of advanced immunological profiling, the study aspires to uncover key mechanisms that drive the initiation, progression, and complications of autoimmune rheumatic diseases. These analyses will combine single nucleotide polymorphisms (SNP) arrays, multiplex assays, transcriptomics, and flow cytometry staining of peripheral blood mononuclear cells to delineate the interplay between hematopoietic mutations and immune dysregulation.

A further objective is the development of a multimodal framework for disease-specific characterization, enabling precise mapping of mutation-driven phenotypes across diverse autoimmune conditions. This framework will incorporate clinical, molecular, and imaging data.

Additionally, the AYLo study aims to explore the potential role of mLOY and other hematopoietic mutations as biomarkers for disease stratification, prognosis, and therapeutic response. The findings may open avenues for personalized treatment approaches, leveraging the molecular insights to inform targeted interventions and improve patient outcomes in autoimmune rheumatic disorders.

By integrating translational and basic science approaches, this study has the potential to redefine current paradigms in autoimmune disease research and therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male
* > 50 years
* Diagnosis of arthritis (RA, PsA), collagen diseases (SLE, systemic sclerosis, Sjögren's syndrome, mixed connective tissue diseases), vasculitis (eGPA, GPA, MPA, IgG4-related disease, GCA, PMR), sarcoidosis, COPD, ILD or asthma bronchiale confirmed by the treating physician.

Exclusion Criteria:

* Female
* < 50 years

Inclusion Criteria (Healthy controls):

* Male
* > 50 years

Exclusion Criteria (Healthy controls):

* Female
* < 50 years
* autoimmune, rheumatological diease
* pulmonary precondition

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients with XY chromosomes.
Study Population: The study population includes male participants aged 50 years or older, divided into two groups: individuals with specific medical conditions (cases) and healthy controls.
  1. Participants must have a diagnosis confirmed by the treating physician of one or more of the following conditions:
     Arthritis (RA, PsA), CTD (e.g., systemic lupus erythematosus [SLE], systemic sclerosis, Sjögren's syndrome, mixed connective tissue diseases), vasculitis ( eosinophilic granulomatosis with polyangiitis [eGPA], granulomatosis with polyangiitis [GPA], microscopic polyangiitis [MPA], IgG4-related disease, GCA + PMR), sarcoidosis, COPD, ILD, asthma bronchial
  2. Healthy Controls: Healthy male participants aged 50 years or older without any of the following conditions:
     Autoimmune or rheumatological diseases Pulmonary preconditions
  3. Exclusion Criteria:
  For both groups, females and individuals younger than 50 years are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Quantification of the fraction of hematopoietic cells exhibiting mLOY. | Cross sectional. Newly diagnosed patients: At baseline and 12 months after diagnosis).
  Detection and quantification of the fraction of hematopoietic cells exhibiting mLOY in peripheral blood using SNP. Unit of Measure: Percentage (%).

SECONDARY OUTCOMES:
Changes in Immune Cell Phenotype | Cross sectional. Newly diagnosed patients: At baseline and 12 months after diagnosis
  Identification and quantification of immune cell subtypes, using flow cytometry.
  Unit of Measure: Changes in levels (percentages).
Changes in Cytokine Profiles | Cross sectional. Newly diagnosed patients: At baseline and 12 months after diagnosis
  Identification and quantification of cytokines using 3'-mRNA transcriptome analysis and ELISA/ Legendplex. Unit of Measure: Changes in levels (pg/mL)
Number of Participants with Detected Pulmonary Involvement | Cross sectional. Newly diagnosed patients: At baseline and 12 months after diagnosis
  Detection of structural anomalies in the lung in clinical routine assessment using lung ultrasound, computed tomography, chest radiography and whole-body plethysmography. Unit of Measure: Number of participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rheumatology, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request from the corresponding author.